CLINICAL TRIAL: NCT07233096
Title: Evaluation of Postoperative Analgesic Efficacy of Ultrasound-Guided Rectus-Intercostal Fascial Plane Block in Living Liver Donors
Brief Title: Rectus-Intercostal Fascial Plane Block for Liver Transplantation Donors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: anestezi 6
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-11

CONDITIONS: Liver Transplantation; Living Donor; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rectus Intercostal Plane Block Group (Active Comparator): Rectus Intercostal Plane Block Group The patients in the Rectus Intercostal Plane Block group will receive a bilateral rectus intercostal plane block and patient-controlled analgesia (PCA) with morphine for postoperative analgesia.
  Interventions: Other: Rectus Intercostal Plane Block
- Control Group (Active Comparator): The patients in the Control group will not receive any regional block and will receive PCA with morphine for postoperative analgesia.
  Interventions: Other: Control (No Block)

INTERVENTIONS:
Other: Rectus Intercostal Plane Block — Rectus intercostal plane block will be administered bilaterally at the end of the surgery and after skin closure under ultrasound guidance
  Arms: Rectus Intercostal Plane Block Group
Other: Control (No Block) — Ultrasound probe placement on the same region without needle insertion or local anesthetic injection to maintain blinding.
  Arms: Control Group

SUMMARY:
Postoperative pain control plays a crucial role in enhancing recovery and improving early mobilization in living liver donors. The rectus-intercostal fascial plane (RIFP) block is a novel ultrasound-guided regional anesthesia technique that provides anterior abdominal wall analgesia by targeting the intercostal nerves between the rectus abdominis and intercostal muscle fascia.

This prospective, randomized controlled clinical study aims to evaluate the postoperative analgesic efficacy and opioid-sparing effects of the RIFP block compared with standard intravenous analgesia in living liver donors undergoing donor hepatectomy.

Participants will be randomly assigned to two groups:

Group 1 (RIFP Block): Patients receiving an ultrasound-guided rectus-intercostal fascial plane block using 20 mL of 0.25% bupivacaine at the end of surgery, in addition to standard IV PCA (morphine).

Group 2 (Control): Patients receiving only standard IV PCA (morphine) without regional block.

DETAILED DESCRIPTION:
This prospective randomized controlled study will include living liver donors undergoing donor hepatectomy. Participants will be divided into two groups: the Rectus-Intercostal Fascial Plane (RIFP) Block Group and the Control Group.

In the RIFP group, patients will receive an ultrasound-guided RIFP block at the end of surgery and postoperative analgesia with intravenous morphine PCA. The control group will receive only intravenous morphine PCA without any regional block.

The primary outcome is total morphine consumption during the first 24 postoperative hours.

Secondary outcomes include pain scores at 1, 6, 12, and 24 hours, time to first rescue analgesia, amount of rescue analgesic used, and incidence of postoperative nausea and vomiting.

This study aims to evaluate the postoperative analgesic efficacy and opioid-sparing effect of the RIFP block in living liver donors compared with standard intravenous analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Patients with American Society of Anesthesiology (ASA) physical status I-II
* Patients scheduled for a living donor hepatectomy

Exclusion Criteria:

* Allergy to local anesthetics
* Coagulopathy
* Skin infection at the block area
* Advanced renal failure
* Chronic pain syndromes
* Alcohol or drug abuse
* Psychiatric disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption | Postoperative 24 hours
  The amount of morphine required by the patient and given by the device will be recorded for the first 24 hours.

SECONDARY OUTCOMES:
Postoperative visual analog scale scores | Postoperative 24 hours
  Postoperative pain will be assessed using a visual analog scale (VAS) (from 0 = no pain to 10 = maximum possible pain) for the first 24 hours.
Rescue analgesic drug consumption | postoperative 24 hours
  The amount of rescue analgesic in mg required by the patient will be recorded for the first 24 hours.
Incidence of postoperative nausea and vomiting | postoperative 24 hours
  Number of patients developing postoperative nausea and vomiting will be recorded for the first 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- istinye University, Istanbul, Turkey (Türkiye)